CLINICAL TRIAL: NCT01728701
Title: Controlled Human Malaria Infection (CHMI) After Immunization With Cryopreserved Plasmodium Falciparum Sporozoites Under Chloroquine Prophylaxis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TIP5; 2012-000322-21 (EudraCT Number)
Record Dates: First submitted 2012-11-06; First posted 2012-11-20 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2014-05

CONDITIONS: Malaria; Plasmodium Falciparum
Keywords: Malaria; Plasmodium falciparum; PfSPZ Challenge; Chemoprophylaxis; PfSPZ-CVac
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Grp 1: 75,000 PfSPZ Challenge, 3 immunizations (Experimental): Grp 1 (10 volunteers) receive std weekly chloroquine (CQ) chemoprophylaxis for 14 weeks(98 days). In this time, Grp 1 gets 6 ID injections of PfSPZ Challenge (total 75,000 PfSPZ NF54 strain), on days 8, 36 & 64 (immunizations 1, 2 & 3). 33 days after last dose of CQ, Grp 1 will have CHMI by bites of 5 mosquitoes infected with Pf NF54 strain.
  Interventions: Biological: PfSPZ Challenge
- Grp 2: Normal Saline (NS) (Placebo Comparator): Grp 2 (5 volunteers) receive std weekly chloroquine (CQ) chemoprophylaxis for 14 weeks(98 days). In this time, Grp 2 gets ID injections of normal saline, on days 8, 36 & 64 (immunizations 1, 2 & 3). 33 days after last dose of CQ, Grp 2 will have CHMI by bites of 5 mosquitoes infected with Pf NF54 strain.
  Interventions: Biological: Normal Saline (NS)
- Grp 3: 75,000 PfSPZ Challenge, 3/4 immunizations (Experimental): Grp 3 (10 volunteers) receive std weekly chloroquine (CQ) chemoprophylaxis for 14 weeks(98 days). In this time, Grp 3 gets 6 ID injections of PfSPZ Challenge (total 75,000 PfSPZ NF54 strain), on days 8, 36 & 64 (immunizations 1, 2 & 3). Grp 3 outcome is dependent on results of Grp 1. If ≥75% of Grp 1 are protected against homologous Pf CHMI, Grp 3 will have CHMI by bites of 5 mosquitoes infected with heterologous Pf NF135.C10 strain 75 days after last dose of CQ. If <75% of Grp 1 are protected against homologous Pf CHMI, Grp 3 will receive 1 additional immunization (immunization 4), consisting of 6 ID injections on the same day of 75,000 PfSPZ Challenge, at day 162. In this 4th immunization period CQ will be administered for another 6 weeks starting at day 154. Finally, 33 days after last dose of CQ, Grp 3 will have homologous Pf CHMI by bites of 5 PfSPZ-infected mosquitoes.
  Interventions: Biological: PfSPZ Challenge
- Grp 4: Normal Saline (NS) (Placebo Comparator): Grp 4 (5 volunteers) receive std weekly chloroquine (CQ) chemoprophylaxis for 14 wks(98 days). In this time, Grp 4 gets ID injections of NS, on days 8, 36 & 64 (immunizations 1, 2 & 3). Grp 4 outcome is dependent on results of Grp 1. If ≥75% of Grp 1 are protected against homologous Pf CHMI, Grp 4 will have CHMI by bites of 5 mosquitoes infected with heterologous Pf NF135.C10 strain 75 days after last dose of CQ. If <75% of Grp 1 are protected against homologous Pf CHMI, Grp 4 will receive 1 additional immunization (immunization 4), consisting of ID injections of NS, at day 162. In this 4th immunization period CQ will be administered for another 6 weeks starting at day 154. Finally, 33 days after last dose of CQ, Grp 4 will have homologous Pf CHMI by bites of 5 PfSPZ-infected mosquitoes.
  Interventions: Biological: Normal Saline (NS)

INTERVENTIONS:
Biological: PfSPZ Challenge — PfSPZ Challenge is a suspension of aseptic, purified, cryopreserved PfSPZ that are thawed and formulated in diluent on the day of administration.
  Arms: Grp 1: 75,000 PfSPZ Challenge, 3 immunizations; Grp 3: 75,000 PfSPZ Challenge, 3/4 immunizations
Biological: Normal Saline (NS) — Normal saline
  Arms: Grp 2: Normal Saline (NS); Grp 4: Normal Saline (NS)

SUMMARY:
The purpose of the study is to determine the safety and tolerability of ID administration of PfSPZ Challenge to volunteers taking chloroquine chemoprophylaxis (an approach called PfSPZ-CVac).

DETAILED DESCRIPTION:
The study is a single centre, double blind, randomized controlled clinical trial. Volunteers, investigators and laboratory personnel will be blinded.

A maximum of 30 volunteers will be randomly divided into four groups. All volunteers will receive standard weekly chloroquine chemoprophylaxis for a period of 14 weeks (98 days). During this period, groups 1 and 3 will receive six ID injections of PfSPZ Challenge, containing a total of 75,000 PfSPZ of the Pf NF54 strain, on days 8, 36 and 64 (immunizations 1, 2 and 3). The control groups 2 and 4 will receive ID injections with normal saline (NS) on the same days.

Thirty-three days after the last dose of chloroquine, volunteers in groups 1 and 2 will have controlled human malaria infection (CHMI) by the bites of five mosquitoes infected with PfSPZ of the Pf NF54 strain. If ≥75% of volunteers in group 1 are protected against this homologous Pf CHMI, volunteers in groups 3 and 4 will have CHMI by the bites of five mosquitoes infected with the heterologous Pf NF135.C10 strain 75 days after the last dose of chloroquine.

If <75% of volunteers in group 1 are protected against the homologous Pf CHMI, volunteers in groups 3 and 4 will receive an additional immunization (immunization 4), which will consist of six ID injections on the same day of 75,000 PfSPZ Challenge and NS respectively, at day 162. In this fourth immunization period chloroquine will be administered for another 6 weeks starting at day 154. Finally, 33 days after the last dose of chloroquine, volunteers in groups 3 and 4 will have homologous Pf CHMI by the bites of five PfSPZ-infected mosquitoes.

After CHMI all volunteers will be treated with a curative regimen of Malarone® (each tablet containing 250 mg atovaquone and 100 mg proguanil), either at the time of detection of blood stage parasitemia or 21 days after exposure to PfSPZ-infected mosquitoes. Volunteers will be checked for parasites by thick smear at least twice after treatment.

If one of the volunteers is not fit to participate in the study on day -1, an alternate volunteer who passed screening will replace him or her. For this purpose 3 additional volunteers will be screened for possible back up.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (males or females) of ≥ 18 and ≤ 35 years of age
* Good health based on history and clinical examination (physical examination and laboratory screening)
* Negative pregnancy test
* Use of adequate contraception for females
* Signing of the informed consent form, thereby demonstrating understanding of the meaning and procedures of the study
* Agreement to inform the general practitioner and to sign a request to release medical information concerning contraindications for participation in the study
* Willingness to undergo administration of PfSPZ Challenge by needle and syringe and willingness to undergo challenge by mosquito bites
* For volunteers not living in Nijmegen: agreement to stay in a hotel room close to the trial centre or living in Nijmegen with a third party that could contact the clinicians in case of alteration of consciousness during a part of the study (day 5 after challenge until treatment is finished)
* Reachable (24/7) by mobile phone during the whole study period
* For volunteers living in Nijmegen: living with a third party that could contact the clinicians in case of alteration of consciousness or agreement to stay in a hotel room close to the trial centre during a part of the study (day 5 after challenge until treatment is finished)
* Available to attend all study visits
* Agreement to refrain from blood donation to Sanquin or for other purposes, during the whole study period
* Willingness to undergo HIV, hepatitis B and hepatitis C tests
* Negative urine toxicology screening test at screening visit and the day before challenge
* Willingness to take a prophylactic regime of chloroquine and a curative regimen of Malarone®
* Willingness to undergo ophthalmologic examination after passing all other inclusion criteria

Exclusion Criteria:

* History of malaria
* Plans to travel to malaria endemic areas during the study period
* Plans to travel outside of the Netherlands during the challenge period
* Previous participation in any malaria vaccine study and/or positive serology for Pf
* Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
* History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
* History of arrhythmias or prolonged QT-interval
* Positive family history of 1st and/or 2nd degree relatives who experienced cardiac events when < 50 years old
* An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
* Clinically significant abnormalities in electrocardiogram (ECG) at screening
* Body Mass Index (BMI) below 18 or above 30 kg/m2
* Any clinically significant deviation from the normal range in biochemistry or haematology blood tests
* Positive HIV, HBV or HCV tests
* Participation in any other clinical study within 30 days prior to the onset of the study
* Enrolment in any other clinical study during the study period
* For women: pregnancy or lactation
* Volunteers unable to give written informed consent
* Volunteers unable to be closely followed for social, geographic or psychological reasons
* History of drug or alcohol abuse interfering with normal social function during a period of one year prior to enrolment in the study
* A history of psychiatric disease
* A history of convulsions
* Known hypersensitivity to Malarone® or chloroquine
* The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids are allowed) and during the study period
* Contraindications to Malarone® or chloroquine including treatment taken by the volunteer that interferes with Malarone® or chloroquine
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia
* Co-workers or trainees of the departments of Medical Microbiology or Internal Medicine of the RUNMC
* Known history of sickle cell anaemia, sickle cell trait, thalassemia, thalassemia trait or G6PD deficiency. If there is any suspicion of G6PD deficiency (based on medical history during screening or ethnic background -Mediterranean, African, or Asian), we will assess G6PD status of that particular subject before inclusion.
* Abnormalities during ophthalmologic examination

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Frequency and magnitude of adverse events in study groups | All study visits+as reported by volunteer upto 53 weeks
  Signs and symptoms will be recorded at all visits, and whenever a trial volunteer reports signs or symptoms to the trial physician between visits. The following signs and symptoms will be solicited: Fever, Headache, Malaise, Fatigue, Dizziness, Myalgia, Arthralgia, Nausea, Vomiting, Chills, Diarrhoea, Abdominal pain (Verhage 2005), Chest pain, Palpitations and Shortness of breath.

SECONDARY OUTCOMES:
Presence of parasitemia after Pf CHMI as assessed by microscopy | Thick smears will be performed on all visits following immunizations and Pf CHMI until treatment is finished upto 53 weeks
  Thick smear samples will be taken from a 3 ml EDTA vacutainer tube. Thick smears will be performed on all visits following immunizations and Pf CHMI until treatment is finished.
  Thick smears will be performed according to a standard operating procedure, which is based on an internationally harmonized protocol for thick smears in CHMIs (Moorthy et al., WHO). In short, 15μl of whole blood will be distributed on standardized 3-well slides, providing an equal slide thickness for all smears. Slides are dried and stained with Giemsa. Per slide, 200 fields will be read, which correlates to 0.5 µl of blood. Slides are considered positive if they contain 2 or more parasites per 200 fields. Thick smears evaluation will take place at the RUNMC.
Time to parasitemia after Pf CHMI as assessed by microscopy | Thick smears will be performed on all visits following immunizations and Pf CHMI until treatment is finished upto 53 weeks
  Thick smear samples will be taken from a 3 ml EDTA vacutainer tube. Thick smears will be performed on all visits following immunizations and Pf CHMI until treatment is finished.
  Thick smears will be performed according to a standard operating procedure, which is based on an internationally harmonized protocol for thick smears in CHMIs (Moorthy et al., WHO). In short, 15μl of whole blood will be distributed on standardized 3-well slides, providing an equal slide thickness for all smears. Slides are dried and stained with Giemsa. Per slide, 200 fields will be read, which correlates to 0.5 µl of blood. Slides are considered positive if they contain 2 or more parasites per 200 fields. Thick smears evaluation will take place at the RUNMC.
Kinetics of parasitemia as assessed by qPCR | Samples collected on all visits following immunizations and Pf CHMI until treatment is finished upto 53 weeks
  Samples for qPCR will be collected from the same 3 ml EDTA vacutainer tubes as the thick smear sample. qPCR will be performed according to standard procedure described in Hermsen et al. Mol, Biochem. Parasitol. 2001; 118: 247-251. In short, qPCR will be performed on the multicopy 18S ribosomal RNA gene. All samples are spiked with murine white blood cells and a murine albumin gene PCR is used to determine efficacy of DNA isolation.
  Samples for quantitative measurement of parasitemia will be prepared and stored at RUNMC. Measurement by qPCR will be performed retrospectively.

OTHER OUTCOMES:
Immune responses in study groups: Cellular immune responses, Antibody production, Cytokine profile | Baseline and throughout the period of study upto 53 weeks
  The overall objective is to find immunological markers or signatures that associate with protective efficacy at immune RNA profile or cell response level.
  Immunogenicity assays will be performed on samples from both vaccinees and infectivity controls from baseline and throughout the period of study.
  Humoral assessment will include antibody assays by immunofluorescence, ELISAs for specific Pf proteins and serological activity with a proteome chip representing thousands of Pf proteins. In addition antibody functionality will be tested in a series of sporozoite inhibition assays.
  Cellular assessment of parasite-specific (subset)T cell responses, will be conducted by multi-parameter flow cytometry and ELISPOT assays) using Pf-specific in vitro stimulation by a number of antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sauerwein, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands